CLINICAL TRIAL: NCT05954728
Title: Cognitive and Neural Mechanisms of Cognitive-behavioral Therapy for Avoidant/Restrictive Food Intake Disorder
Brief Title: Cognitive-behavioral Therapy vs. Nutrition Counseling for Avoidant/Restrictive Food Intake Disorder
Acronym: COUNTERACT
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Jennifer Thomas, Eating Disorder Clinical and Research Program (EDCRP) Co-Director/Associate Professor of Psychiatry, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023P001491
Record Dates: First submitted 2023-07-05; First posted 2023-07-20 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Avoidant/Restrictive Food Intake Disorder (ARFID)
MeSH Terms: conditions — Avoidant Restrictive Food Intake Disorder | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CBT-AR (Experimental): See intervention description
  Interventions: Behavioral: Cognitive-Behavioral Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR)
- Nutrition Counseling (Experimental): See intervention description
  Interventions: Behavioral: Nutrition Counseling for Avoidant/Restrictive Food Intake Disorder

INTERVENTIONS:
Behavioral: Cognitive-Behavioral Therapy for Avoidant/Restrictive Food Intake Disorder (CBT-AR) — CBT-AR is a four-stage modular treatment for ARFID delivered by a mental health clinician. The four stages include: 1) Psychoeducation and early change; 2) Treatment planning; 3) Addressing maintaining mechanisms; and 4) Relapse prevention. For participants ages 10-15 years, patients/guardians attend the sessions. For patients ages 16 and up, the therapy is individual.
  Arms: CBT-AR
Behavioral: Nutrition Counseling for Avoidant/Restrictive Food Intake Disorder — Nutrition counseling will be provided by skilled registered dietitians at the MGH Translational and Clinical Research Center (TCRC). Sessions focus on the foods necessary for a healthy diet, how to meet nutritional needs, how to incorporate healthy exercise, and support for making these changes. For participants ages 10-15 years, patients/guardians attend the sessions. For patients ages 16 and up, the therapy is individual.
  Arms: Nutrition Counseling

SUMMARY:
This study is a randomized controlledlinical trial, assessing the efficacy of cognitive- behavioral therapy (CBT-AR) and nutrition counseling for avoidant/restrictive food intake disorder (ARFID) for children and adolescents (ages 10-18 years).

ELIGIBILITY:
Inclusion Criteria:

* Males and Females ages 10-18 years old
* Current ARFID
* Normal TSH or free T4 levels to rule out thyroid disease as cause of symptoms
* Negative celiac screening panel indicating no active celiac disease as cause of symptoms
* Fluency and literacy in English

Exclusion Criteria:

* BMI < 5th percentile for sex and age
* Pregnancy, breastfeeding, or recent initiation/cessation of oral contraceptive pills within 8 weeks of the pre-treatment study visit
* Current/history of psychosis
* Substance/alcohol use disorder (active within the past month)
* Medical instability requiring inpatient care according to the American Psychiatric Association 2023 treatment guidelines for eating disorders
* Laboratory abnormalities indicating a need for higher level of care
* Complete lack of oral intake (suggesting a need for inpatient care)
* Tube feeding (suggesting a need for tube weaning)
* Active suicidal/homicidal ideation with intent or plan
* Contraindications to MRI
* History of major gastrointestinal tract surgery or serious medical condition (e.g., cancer)
* Medical history of intellectual disability
* Illiteracy

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-01-31 (Actual); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Food Neophobia Scale | Change from baseline food neophobia measured at pre-treatment to after each weekly session of treatment and after the complete 15 weeks of treatment measured at post-treatment
  Validated 6-item version of the Food Neophobia Scale used to assess food neophobia on a scale from 1 to 7, with higher scores indicating higher levels of food neophobia. The lowest score possible is 7, indicating low food neophobia, and highest score possible is 42, indicating high food neophobia.
Functional magnetic resonance imaging (fMRI) food cue paradigm | Change from baseline neural activation in response to food cues measured at pre-treatment to after 15 weeks of treatment measured at post-treatment
  Used to measure neural activation in response to food cues. Higher scores indicate higher neural activation. There is no minimum or maximum for this measure.

SECONDARY OUTCOMES:
General Nutrition Knowledge Questionnaire (GNKQ) | Change from baseline measured at pre-treatment to after 15 weeks of treatment measured at post-treatment
  A revised version of the General Nutrition Knowledge Questionnaire (GNKQ) used to evaluate knowledge of nutrition. Scores are gathered through a series of multiple-choice questions. The lowest score possible is 0, indicating low knowledge of nutrition, and the highest score possible is 14, indicating high knowledge of nutrition.
Pica, ARFID, and Rumination Disorder Interview (PARDI) | Change from baseline measured at pre-treatment to after 15 weeks of treatment measured at post-treatment
  A semi-structured clinical interview assessing the symptoms and severity of Pica, ARFID, and Rumination Disorder. This interview is used to determine the presence and severity of each ARFID profile. Scores for each severity measure are assessed on a scale from 0 to 6, with higher scores indicating greater severity.
Pica, ARFID, and Rumination Disorder ARFID Questionnaire (PARDI-AR-Q) | Change from baseline measured at pre-treatment to after 15 weeks of treatment measured at post-treatment
  A 32-item revised version of the Pica, ARFID, and Rumination Disorder Interview used to assess ARFID severity and presence of Pica or Rumination Disorder. Each item is assessed on a scale from 0 to 6, with higher scores indicating greater severity.
4-Day Food Record measuring percent of calories consumed from fruits, vegetables, proteins, grains, and dairy food groups. | Change from baseline measured at pre-treatment to after 15 weeks of treatment measured at post-treatment
  A record of participant diet for four days prior to the Pre-Treatment Assessment and for another four days prior to the Post-Treatment Assessment. Dietary information is calculated from the recorded foods.
24-Hour Recall measuring percent of calories consumed from fruits, vegetables, proteins, grains, and dairy food groups. | Change from baseline measured at pre-treatment to after 15 weeks of treatment measured at post-treatment
  A detailed recall of everything a participant has consumed during the 24 hours prior to the Pre-Treatment Assessment, and again prior to the Post-Treatment Assessment. Dietary information is calculated from the recorded foods.

CONTACTS AND LOCATIONS:
Locations (1):
- Eating Disorders Clinical and Research Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will upload de-identified data to the NIMH National Data Archive at the conclusion of the study